CLINICAL TRIAL: NCT06218771
Title: A Phase Ib Clinical Trial of TQB3454 Tablets in Patients With Blood Tumors
Brief Title: A Study of TQB3454 Tablets in Patients With Blood Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3454-Ib-01
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3454 Tablets (Experimental): TQB3454 Tablets, orally administered, 28 days as a treatment cycle.
  Interventions: Drug: TQB3454 Tablets

INTERVENTIONS:
Drug: TQB3454 Tablets — TQB3454 Tablets is a selective isocitrate dehydrogenase 1 (IDH1) mutation inhibitor

SUMMARY:
The purpose of this clinical trial is to evaluate the safety of TQB3454 tablets in patients with acute myeloid leukemia and myelodysplastic syndrome, and determine the phase II recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily joined the study and signed informed consent with good compliance.
* Men and women; The expected survival is ≥3 months.
* Negative serum/urine pregnancy test within 7 days prior to initial dose and must be non-lactating; Women of childbearing age agree to use contraception (such as an intrauterine device, birth control pill or condom) during the study and for six months after the study completion; Men agreed to use contraception during the study period and for six months after the end of the study.
* The major organs are functioning well;
* For Relapsing/refractory acute myeloid leukemia (AML):

  1. According to the classification criteria for Hematopoietic and lymphoid tissue tumors revised by the World Health Organization (WHO) in 2016, AML confirmed by bone marrow cell morphology, excluding acute promyelocytic leukemia (APL).
  2. ≥18 years old; Eastern Cooperative Oncology Group (ECOG) score is 0~2.
  3. Blood biochemical examination:

  i: Total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN), liver infiltration ≤3×ULN in Gilbert syndrome patients or tumor diseases; ii: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; ALT and AST≤5×ULN if liver infiltration was associated.
* For myelodysplastic syndrome (MDS) with higher risk:

  1. MDS patients were confirmed by bone marrow cell morphology and cytogenetics and met the classification criteria of hematopoietic and lymphoid tissue tumors revised by WHO in 2016.
  2. ≥18 years old; ECOG score is 0~2. c. Blood biochemical examination:

  i: Total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN), liver infiltration ≤3×ULN in Gilbert syndrome patients or tumor diseases.

ii: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; ALT and AST≤5×ULN if concomitant with liver infiltration.

Exclusion Criteria:

* Tumor diseases and history:

  1. The tumor has or is suspected to involve the central nervous system, or primary Central nervous system leukemia.
  2. Present or present with other malignant tumors within 3 years prior to the first dose. Except the following conditions: for other malignancies treated with a single operation, achieving a 5-year continuous disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)].
  3. Severe life-threatening complications of leukemia, such as uncontrolled bleeding, hypoxia or shock pneumonia, and disseminated intravascular coagulation.
* Previous antitumor therapy:

  1. Received National Medical Products Administration (NMPA) approved Chinese patent drugs with anticancer indications specified in the drug label within 2 weeks prior to initial administration.
  2. Toxicities associated with previous antineoplastic therapy did not return to CTCAE≤1, except for hair loss, fatigue and poor appetite.

     3. Associated diseases and history:

  <!-- -->

  1. Abnormal liver.
  2. Renal abnormalities.
  3. Gastrointestinal abnormalities.
  4. Cardio-cerebrovascular abnormalities.
  5. Immune-related history.
  6. Lung disease.
  7. Comorbidities that were severe or poorly controlled and, in the investigator's judgment, significantly compromised patient safety or hindered study completion.
  8. Risk of bleeding.
* History of drug abuse or drug abuse.
* Participated in clinical trials of other drugs within the past 30 days;
* It is estimated that the patient's compliance to participate in this clinical study is insufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The rate of all adverse events (AEs), serious adverse events (SAEs) | Up to 80 weeks
  Proportion of patients with adverse events/serious adverse events, as defined by Common Terminology Criteria for Adverse Events (CTCAE5.0)
The severity of all adverse events (AEs), serious adverse events (SAEs) | Up to 80 weeks
  The severity of adverse events/serious adverse events, as defined by Common Terminology Criteria for Adverse Events (CTCAE5.0)
Incidence of abnormal laboratory values | Up to 80 weeks
  The proportion of patients with abnormal laboratory examination indicators mainly included blood routine, blood routine, blood biochemistry, coagulation function, thyroid function, myocardial enzyme profile, urine routine, stool routine and 12-lead electrocardiogram.

SECONDARY OUTCOMES:
Peak time (Tmax) | Cohort 1: pre-dose on Day 1, 14, 28 of Cycle 1, Day 14, 28 of Cycle 2. 2, 3, 4, 10, 24 hours after dose on Cycle1 Day28. Cohort 2: pre-dose, 2, 3, 4, 10, 24 hours after dose on Day 1, 28 of Cycle 1. Pre-dose on Day 14, 28 of Cycle2. 28 days as a cycle.
  The time required to reach peak concentration after administration.
Peak concentration (Cmax) | Cohort 1: pre-dose on Day 1, 14, 28 of Cycle 1, Day 14, 28 of Cycle 2. 2, 3, 4, 10, 24 hours after dose on Cycle1 Day28. Cohort 2: pre-dose, 2, 3, 4, 10, 24 hours after dose on Day 1, 28 of Cycle 1. Pre-dose on Day 14, 28 of Cycle2. 28 days as a cycle.
  the maximum plasma concentration of the drug after administration.
Area under blood concentration-time curve (AUC 0-24h) | Cohort 1: pre-dose on Day 1, 14, 28 of Cycle 1, Day 14, 28 of Cycle 2. 2, 3, 4, 10, 24 hours after dose on Cycle1 Day28. Cohort 2: pre-dose, 2, 3, 4, 10, 24 hours after dose on Day 1, 28 of Cycle 1. Pre-dose on Day 14, 28 of Cycle2. 28 days as a cycle.
  The area surrounded by the blood concentration curve to the time axis.
Steady-state apparent volume of distribution (Vz/F) | Cohort 1: pre-dose on Day 1, 14, 28 of Cycle 1, Day 14, 28 of Cycle 2. 2, 3, 4, 10, 24 hours after dose on Cycle1 Day28. Cohort 2: pre-dose, 2, 3, 4, 10, 24 hours after dose on Day 1, 28 of Cycle 1. Pre-dose on Day 14, 28 of Cycle2. 28 days as a cycle.
  The volume of distribution at steady-state concentration.
Steady-state blood trough concentration (Cmin,ss) | Cohort 1: pre-dose on Day 1, 14, 28 of Cycle 1, Day 14, 28 of Cycle 2. 2, 3, 4, 10, 24 hours after dose on Cycle1 Day28. Cohort 2: pre-dose, 2, 3, 4, 10, 24 hours after dose on Day 1, 28 of Cycle 1. Pre-dose on Day 14, 28 of Cycle2. 28 days as a cycle.
  the lowest concentration during dosing and is usually obtained from the initial moment after dosing to the lowest concentration before the next dosing when multiple dosing reaches steady-state.
Complete response (CR) rate | Up to 80 weeks
  The proportion of patients with an optimal response of CR.
Complete response (CR) + Complete response with partial hematological recovery (CRh) | Up to 80 weeks
  Proportion of patients with optimal response of CR and CRh
Transfusion-independent improvement | Up to 80 weeks
  Proportion of transfusion-dependent patients at baseline who were removed from red blood cell (RBC) or platelet transfusion dependence after randomization.
CR+CRh duration | Up to 80 weeks
  In all patients with an optimal response of CR or CRh, the time from the date when CR or CRh was first achieved to the date of first clearly documented disease progression / relapse / treatment failure or death, whichever occurs first.
CR duration | Up to 80 weeks
  For all patients with an optimal response of CR, the time from the date when CR was first achieved to the first clearly documented date of disease progression/relapse/treatment failure or death, whichever occurs first.
Duration of response (DOR) | Up to 80 weeks
  The time from the date of first remission to the date of first clearly documented disease progression/relapse/treatment failure or date of death in all patients with optimal response of CR, CR with incomplete blood count recovery(CRi), CR with incomplete platelet recovery (CRp), Morphologic Leukemia-free state (MLFS), or Partial Remission (PR), whichever occurs first.
Time to CR+CRh | Up to 80 weeks
  Time from the date of first TQB3454 dose to the date of first CR or CRh in all patients with optimal response to CR or CRh.
Event-free survival (EFS) | Up to 80 weeks
  The time from the date of the first dose TQB3454 tablet to the first clearly documented date of relapse after disease remission, disease progression/treatment failure, or death, whichever occurs first.
Overall survival (OS) | Up to 80 weeks
  Time from the date of first dose of TQB3454 tablet to the date of death from any cause.
Functional Assessment of Chronic Illness (FACIT) fatigue Scale | Up to 80 weeks
  Proportion of patients with a confirmed improvement of at least 3 points from baseline in FACit-Fatigue scale scores.
Quality of life score | Up to 80 weeks
  Proportion of patients with a confirmed improvement of at least 10 points from baseline in their overall health as assessed by European organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).
Overall response rate (ORR) | Up to 80 weeks
  Proportion of patients with an optimal response of CR, marrow CR (mCR), PR, or Hematology improvement (HI).
Progression-free survival (PFS) | Up to 80 weeks
  from the date of first dose of TQB3454 tablet to the time of first recorded disease progression assessed by the investigator or relapse after CR or death from any cause. Disease progression includes acute leukaemia transformation.
Leukemia-free survival | Up to 80 weeks
  from the date of first dose of TQB3454 tablet to the time of >20% original cells in bone marrow/peripheral blood, or diagnosis of acute extramedullary leukemia, or death from any cause.
Correlation between 2-hydroxyglutaric acid (2-HG) and efficacy | Pre-dose (baseline). Pre-dose on Cycle 1 Day 14, Cycle 1 Day 28, Cycle 2 Day 28, Cycle 3 Day 28, Cycle 4 Day 28, Cycle 5 Day 28, Cycle 6 Day 28, 28 days as a cycle
  Liquid chromatography-mass spectrometry (LC-MS/MS) was used to determine 2-HG in plasma and to analyze its correlation with efficacy.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cangzhou people's Hospital, Cangzhou, Hebei
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Yantai Mountain Hospital, Yantai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality